CLINICAL TRIAL: NCT01203644
Title: A Phase 2, Multicenter, Randomized, Double Blind, Dose Escalating/ De Escalating Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of a Single Dose of Sustained Release Encapsulated Bupivacaine (SKY0402) in the Management of Postoperative Pain in Subjects Undergoing Inguinal Hernia Repair
Brief Title: Evaluation of the Safety, Efficacy, and Pharmacokinetics of SKY0402 in Subjects Undergoing Inguinal Hernia Repair
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SKY0402-C-201
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Results first posted 2012-05-14 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Inguinal Hernia
Keywords: Postoperative pain; Analgesia
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacaine HCl (Active Comparator): (e.g., Marcaine with epinephrine 1:200,000) is the reference-listed drug for bupivacaine and contains the same active, local anesthetic as SKY0402
  Interventions: Drug: SKY0402
- SKY0402 (Active Comparator): Low dose, low-mid dose, mid-dose, and high dose
  Interventions: Drug: Bupivacaine HCl

INTERVENTIONS:
Drug: SKY0402 — Single dose of SKY0402 administered locally into the surgical wound.
  Arms: Bupivacaine HCl
Drug: Bupivacaine HCl — Single dose of bupivacaine HCl (100 mg) administered locally into the surgical wound.
  Arms: SKY0402

SUMMARY:
The primary objective of this study was to determine the appropriate dose of SKY0402 for the management of postoperative pain following inguinal hernia repair. This study evaluated the safety, efficacy, and pharmacokinetics of SKY0402 compared with a 100 mg dose of bupivacaine HCl for the treatment of postoperative pain in subjects undergoing inguinal hernia repair. Study drug was administered by surgical wound infiltration at the end of the hernia repair procedure.

DETAILED DESCRIPTION:
SKY0402 was administered in a dose escalating/de-escalating fashion, with a low starting dose in Cohort 1 that was to be increased or decreased in subsequent cohorts based on safety and analgesic effects. The decision to proceed to the next cohort (i.e., increase or decrease the dose) was made by a Cohort Data Review Committee following a review of the data from the previous cohort. Subjects were randomized to receive either SKY0402 or bupivacaine HCl at a ratio of 1:1 in Cohort 1 and at a ratio of 3:1 in subsequent cohorts. The dose of bupivacaine HCl (100 mg) remained constant for all cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Males ≥18 years of age at the Screening visit.
2. Scheduled to undergo unilateral inguinal hernia repair under general anesthesia, using an open, tension free procedure (e.g., Lichtenstein technique with or without mesh).
3. American Society of Anesthesiology (ASA) Physical Class 1 or 2.
4. Able and willing to comply with all study visits and procedures.
5. Capable of speaking and understanding the local language sufficiently to provide responses to pain assessment scales.
6. Willing and capable of providing written informed consent.

Exclusion Criteria:

1. Clinically significant electrocardiogram abnormalities at Screening or on Day 1 (pre administration).
2. Albumin and/or alpha 1 acid glycoprotein (AAG) below normal levels.
3. Current or historical evidence of any clinically significant disease or condition that, in the opinion of the Investigator, might have increased the risk of surgery or complicated the subject's postoperative course.
4. Opioid medication usage during the 7 day period preceding the administration of study drug.
5. Current medical conditions that could have required treatment with analgesic medications in the postoperative period for pain that was not surgically related (e.g., rheumatoid arthritis).
6. Body mass index >30 kg/m^2
7. Body weight <60 kg.
8. History of hypersensitivity or idiosyncratic reaction to amide type local anesthetic agents.
9. History of hypersensitivity, idiosyncratic reactions, and other contraindications to the pain control agents (opioid or non-opioid) anticipated to be used postoperatively. These contraindications may have included: angioedema and bronchospastic reactivity to non steroidal anti inflammatory drug, peptic ulcer (active within the last three months), hepatic or renal insufficiency.
10. Coagulation disorders or ongoing anticoagulation treatment.
11. Administration of an investigational drug within 30 days or five half lives (of elimination), whichever was longer, prior to study drug administration.
12. Suspected or known history of substance abuse and/or alcoholism.
13. Clinically significant complications during the hernia repair surgery (e.g., excessive bleeding), which might have rendered the subject medically unstable or might have complicated the subject's postoperative course.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2004-12; Primary Completion 2006-01 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kay Warnott, RN, ACNP, Study Director — Pacira Pharmaceuticals, Inc

REFERENCES:
- [Derived] Dasta J, Ramamoorthy S, Patou G, Sinatra R. Bupivacaine liposome injectable suspension compared with bupivacaine HCl for the reduction of opioid burden in the postsurgical setting. Curr Med Res Opin. 2012 Oct;28(10):1609-15. doi: 10.1185/03007995.2012.721760. Epub 2012 Sep 3. PMID 22900785

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bupivacaine HCl | SKY0402
Started | 26 | 50
Completed | 26 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine HCl | SKY0402 | Total
Number analyzed (Participants) | 26 | 50 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 36 | 60
  >=65 years | 2 | 14 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (12.6) | 55.1 (16) | 53.8 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 26 | 50 | 76
Region of Enrollment [Number; unit: participants]
  Belgium | 0 | 8 | 8
  Australia | 16 | 26 | 42
  United Kingdom | 4 | 12 | 16
  Netherlands | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Time to First Use of Supplemental Pain Medication
Description: The primary efficacy endpoint was the time to first use of supplemental pain medication (opioid or non-opioid) postoperatively for surgical wound pain
Time Frame: Through 96 hours postdose
Measure: Median (Inter-Quartile Range); unit: hours
Groups:
- Bupivacaine HCl: (e.g., Marcaine with epinephrine 1:200,000) is the reference-listed drug for bupivacaine and contains the same active, local anesthetic as SKY0402. Single 100 mg administration of 0.25% solution (i.e., 0.5% diluted 1:1) in a 40-mL volume via local infiltration
- SKY0402 Low Dose: Single administration of SKY0402 (low dose, 175 mg) in a 40-mL volume via local infiltration
- SKY0402 Low-mid Dose: Single administration of SKY0402 (low-mid dose, 225 mg) in a 40-mL volume via local infiltration
- SKY0402 High-mid Dose: Single administration of SKY0402 (high-mid dose, 300 mg) in a 40-mL volume via local infiltration
- SKY0402 High Dose: Single administration of SKY0402 (high dose, 350 mg) in a 40-mL volume via local infiltration
Arm/Group | Bupivacaine HCl | SKY0402 Low Dose | SKY0402 Low-mid Dose | SKY0402 High-mid Dose | SKY0402 High Dose
Number analyzed (Participants) | 26 | 12 | 12 | 12 | 14
hours | 4.2 [1.3 to 13.7] | 13.75 [2.1 to 62.7] | 3.9 [0.8 to 7.4] | 5.2 [1.9 to 18.8] | 5.5 [1.4 to 96]

2. Secondary Outcome: Adverse Events
Description: Safety assessments included monitoring of treatment-emergent adverse events
Time Frame: Through 30 days postdose
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Bupivacaine HCl | SKY0402
Serious Adverse Events (participants affected / at risk) | 0/26 | 2/50
Other Adverse Events (participants affected / at risk) | 10/26 | 12/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bupivacaine HCl (N=26) | SKY0402 (N=50)
Postoperative hematoma (Injury, poisoning and procedural complications) | 0 | 1 — Occurred in the low-mid dose group
Urinary Retention/BPH (Renal and urinary disorders) | 0 | 1 — Occurred in the high-mid dose group
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bupivacaine HCl (N=26) | SKY0402 (N=50)
Nausea (Gastrointestinal disorders) | 2 | 4
Localized oedema (General disorders) | 2 | 1
Pyrexia (General disorders) | 1 | 3
Wound infection (Infections and infestations) | 2 | 0
Urinary retention (Renal and urinary disorders) | 2 | 1
Hypertension NOS (Vascular disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No